CLINICAL TRIAL: NCT05003843
Title: BOLT: A Prospective, Multicenter Study of Patients With Deep Vein Thrombosis to Evaluate the Safety and Efficacy of the Indigo® Aspiration System
Brief Title: BOLT: Study of the Indigo® Aspiration System When Used in Patients With Deep Vein Thrombosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19458
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Deep Vein Thrombosis; DVT
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Other): Use of Indigo Aspiration System in patients with obstruction due to DVT
  Interventions: Device: Indigo Aspiration System

INTERVENTIONS:
Device: Indigo Aspiration System — Indigo Aspiration System

SUMMARY:
The objective of this study is to demonstrate the safety and efficacy of the Indigo Aspiration system for percutaneous mechanical thrombectomy in a population presenting with obstruction due to deep vein thrombosis (DVT) who are eligible for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral lower extremity DVT occlusion involving iliac and/or common femoral veins with up to 2 cm extension in the inferior vena cava (IVC) or femoral in combination with iliac veins, including patients with extension of clot into the contralateral common iliac vein Note: Patients with non-iliofemoral DVT in the contralateral limb, who do not require endovascular treatment, may be enrolled
* Acute thrombotic or thromboembolic occlusion with symptom duration of 14 days or less at presentation
* Frontline treatment with Indigo Aspiration System in the target venous segment per Investigator decision
* Patient is ≥18 years of age
* Informed consent is obtained per Institutional Review Board requirements

Exclusion Criteria:

* Contraindication to systemic or therapeutic doses of anticoagulants
* Contraindication to iodinated contrast venography that cannot be adequately premedicated
* Complete infrarenal IVC occlusion
* In the index leg: prior DVT
* Prior stent in target venous segment
* Treatment of index DVT with thrombolytics within 14 days prior to index procedure
* Pulmonary embolism (PE) defined as either high (systolic blood pressure < 90 mmHg and/or patient on IV vasoactive medication to support blood pressure), or intermediate high-risk PE, as defined by the European Society Guideline on management of PE. Low risk PE and/or intermediate low risk PE can be enrolled.
* Known coagulation disorders both acquired (e.g., Heparin Induced Thrombocytopenia, etc.) or genetic (e.g., Factor V Leiden, etc.), thrombophilia, or hypercoagulable state
* Pregnant patients
* Life expectancy <1 year due to comorbidities
* Primary brain, metastatic cancer or marrow malignancies
* Current participation in another investigational drug or device study that may confound the results of this study. Studies requiring extended follow-up for products that were investigational but have since become commercially available are not considered investigational studies.
* Other medical, behavioral, or psychological conditions that, in the opinion of the Investigator, precludes the patient from appropriate consent, could limit the patient's ability to participate in the study, including compliance with follow-up requirements, or that could impact the scientific integrity of the study
* Pre-existing malpositioned stent(s) that obstructs the ostium of the index iliac vein and contacts the vena cava wall as demonstrated by venography prior to the index procedure
* Congenital anatomic anomalies of the IVC or iliac veins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-11-18 (Actual); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Composite of Major Adverse Events | 48 Hours Post-Procedure
  Device related death, major bleeding, new symptomatic pulmonary embolism or re-thrombosis of the target venous segment and serious device related events
Change in Marder Score | Index Procedure
  Complete or near complete (75% or greater) reduction of venous thrombus from the target venous segment as measured by Marder Score pre- to post-procedure
  The Marder Score ranges from 0 to 24, with higher scores being worse.

SECONDARY OUTCOMES:
Composite of Major Adverse Events | 30 Days Post-Procedure
  A composite of death, major bleeding, new symptomatic pulmonary embolism or re-thrombus of the target venous segment
Device Related Adverse Events | 24 Months
  Proportion of participants with device related adverse events
Villalta Scale | 24 Months
  Villalta scores reported at baseline, 30 days, 180 days, 12 months, and 24 months
  Villalta score ranges from 0 (no post thrombotic syndrome) to 33 (severe post thrombotic syndrome), with higher scores being worse.

CONTACTS AND LOCATIONS:
Locations (42):
- United States (42):
  - Sharp Grossmont, La Mesa, California
  - Long Beach Medical Center, Long Beach, California
  - UCLA, Los Angeles, California
  - Christiana Care, Newark, Delaware
  - MedStar Washington, Washington D.C., District of Columbia
  - Memorial Jacksonville, Jacksonville, Florida
  - Radiology and Imaging Specialists, Lakeland, Florida
  - Baptist of Miami, Miami, Florida
  - Mount Sinai Miami, Miami Beach, Florida
  - Sarasota Memorial, Sarasota, Florida
  - Protestant Memorial Medical Center, Inc, Belleville, Illinois
  - Northwestern Memorial, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - St. Vincent, Indianapolis, Indiana
  - Indiana University Health, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Lafayette General/Cardiovascular Institute of the South, Lafayette, Louisiana
  - LSU Hospital Shreveport, Shreveport, Louisiana
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - St. Joseph Mercy Ann Arbor Hospital, Ann Arbor, Michigan
  - McLaren Greater Lansing, East Lansing, Michigan
  - Jewish Barnes Hospital, St Louis, Missouri
  - Nebraska Methodist, Omaha, Nebraska
  - Hackensack Medical Center, Hackensack, New Jersey
  - Lovelace Heart, Albuquerque, New Mexico
  - Kaleida University at Buffalo, Buffalo, New York
  - Weill Cornell Medicine, New York, New York
  - Mount Sinai NY, New York, New York
  - Lenox Hill Hospital, New York, New York
  - NYU, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - Christ Cincinnati, Cincinnati, Ohio
  - TriHealth, Cincinnati, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - UPenn, Philadelphia, Pennsylvania
  - MUSC, Charleston, South Carolina
  - Holston Valley Medical, Kingsport, Tennessee
  - BUMC - Dallas (Scott & White), Dallas, Texas
  - Sentara, Norfolk, Virginia